CLINICAL TRIAL: NCT05270889
Title: An Open Label, Single-Arm, Multi-center Phase II Study to Evaluate the Safety and Efficacy of Tislelizumab in Combination With Zanidatamab as a 2nd Line in HER2-Positive Advanced Gastric Cancer in K-Umbrella Trial
Brief Title: Study to Evaluate the Safety and Efficacy of Tislelizumab in Combination With Zanidatamab as a 2nd Line in HER2-Positive Advanced Gastric Cancer in K-Umbrella Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1475
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: HER2-positive Gastric Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tislelizumab+Zanidatamab (Experimental)
  Interventions: Drug: Tislelizumab+Zanidatamab

INTERVENTIONS:
Drug: Tislelizumab+Zanidatamab — Zanidatamab will be administered at a flat dose as follows:
  * Subjects with body weight <70 kg: 1800 mg IV on Day 1 of each 21-day cycle
  * Subjects with body weight ≥70 kg: 2400 mg IV on Day 1 of each 21-day cycle Tislelizumab will be administered at a dose of 200 mg IV on Day 1 of each cycle.

SUMMARY:
Study Design:

This is a Phase II study to assess the safety and clinical efficacy of this combined chemotherapy-free regimen (zanidatamab and tislelizumab) in HER2-positive advanced gastric/gastroesophageal junction (GEJ) adenocarcinoma after first line treatment. The study will be conducted as phase II study to evaluate the safety and tolerability of the combination treatment of zanidatamab and tislelizumab and determine anti-tumor activity in HER2-positive advanced gastric/GEJ adenocarcinoma patients. This study will be conducted at up to 6 medical centers in Korea. Patients who are HER2-positive will be confirmed by immunohistochemistry (IHC) or fluorescent in situ hybridization (FISH)/silver in situ hybridization (SISH) at local laboratory. Patients who meet all eligibility criteria will be enrolled to this study and receive treatment with zanidatamab and tislelizumab until progressive disease is confirmed or at least 1 discontinuation criterion is met.

Study Assessments:

Patients will be monitored for safety, tolerability, and antitumor activity throughout the study. Safety will be assessed throughout the study by monitoring AEs/SAEs, and laboratory results. Vital signs, physical examinations, Eastern Cooperative Oncology Group (ECOG) performance status change, ECG results, echocardiogram/MUGA, and other examinations will also be used for safety assessment. Anticancer activity will be evaluated by the investigator using RECIST 1.1. Radiological assessment of tumor response status will be performed every 6 weeks (±7 days) from (anchored to) Cycle 1 Day 1 for the first 54 weeks and every 12 weeks (±7 days) thereafter until disease progression, withdrawal of consent, death, or start of a new anticancer therapy.

Patients who discontinue study treatment early for reasons other than disease progression will continue to undergo tumor assessments following the original plan until the patient begins a subsequent anticancer treatment, experiences disease progression, withdraws consent, is lost to follow up, death, or until the study terminates, whichever occurs first.

Duration of Patient Participation:

Screening Period is within 28 days prior to the first dose of study drug. Treatment Period starts with the first dose administration of study drug and ends when the patient is discontinued for study treatment when they are no longer considered to be achieving clinical benefit due to confirmed disease progression or unacceptable toxicity, or due to death or withdrawal of consent.

Safety Follow-up. Patients who discontinue treatment for any reason will be asked to return to the clinic for the Safety Follow up Visit (to occur approximately 30 days (±7 days] after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first). In addition, telephone contacts with patients treated with zanidatamab and tislelizumab should be conducted to assess immune-mediated AEs and concomitant medications (if applicable, i.e. associated with an immune-mediated AE or is a new anticancer therapy) at 60 (±14 days) and 90 days (±14 days) after the last dose of study drug(s) regardless of whether the patient starts a new anticancer therapy.

Survival Follow-up. Patients will be followed for survival and further anticancer therapy information after discontinuation of study treatment via telephone calls, patient medical records, and/or clinic visits approximately every 3 months (±14 days) after the Safety Follow-up Visit or as directed by the investigator until death, loss to follow-up, withdrawal of consent, or study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Age ≥19 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
3. Has a histologically or cytologically confirmed diagnosis of advanced gastric /GEJ adenocarcinoma (systemic metastasis or locally advanced unresectable gastric/GEJ adenocarcinoma)
4. Progressed from prior 1st line systemic chemotherapy (no more than one previous line of treatment is allowed; trastuzumab or other anti-HER2 therapy is acceptable as prior treatment, except for zanidatamab)
5. Has a documented HER2-positive tumor in primary or metastatic tumor tissue

   1. HER2-positive tumor defined as either IHC 3+; OR
   2. IHC 2+ in combination with SISH + (or FISH), as assessed by local laboratory on primary or metastatic tumor (SISH positivity is defined as a ratio of ≥2.0 for the number of HER2 gene copies to the number of signals for CEP17)
6. Has measurable disease as determined by RECIST 1.1 (A lesion which received prior radiotherapy cannot be a measurable lesion.)
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
8. LVEF ≥50% as determined by either echocardiogram or multiple gated acquisition scan (MUGA)
9. Adequate organ function as indicated by the following laboratory values during screening

   a. Patients must not have required a blood transfusion or growth factor support ≤14 days before sample collection at screening for the following: i. Absolute neutrophil count (ANC) ≥1.5 x 109/L ii. Platelets ≥75 x 109/L iii. Hemoglobin ≥90 g/L b. Serum creatinine ≤1.5 x ULN (upper limit of normal) or estimated Glomerular Filtration Rate ≥60 mL/min/1.73 m2 (Appendix 8) c. Serum total bilirubin ≤1.5 x ULN (total bilirubin must be <3 x ULN for patients with Gilberts syndrome) d. AST and ALT ≤3 x ULN
10. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and for 7 months after the last dose of study drugs, and have a negative urine or serum pregnancy test ≤7 days of first dose of study drug (Appendix 9)
11. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for 7 months after the last dose of study drugs (Appendix 9)
12. Male subjects must agree not to donate sperm and female subjects must agree not to donate oocytes starting at screening and throughout the study period, and for 7 months after treatment discontinuation

Exclusion Criteria:

1. Have previously received zanidatamab (trastuzumab or other anti-HER2 therapy is acceptable as a prior treatment).
2. Have previously received Tislelizumab, anti-programmed cell death-1 (PD-1) antibody, anti-PD-L1 antibody, anti-programmed cell death-ligand 2 (PD-L2) antibody, anti-CD137 antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) antibody, or other therapeutic antibodies or pharmacotherapies for the regulation of T-cells.
3. Active leptomeningeal disease or uncontrolled brain metastasis. Patients with equivocal findings or with confirmed brain metastases are eligible for enrollment provided that they are asymptomatic and radiologically stable without the need for corticosteroid treatment for ≥ 4 weeks before first dose of study drug.

   Note: Eligibility with regards to the anatomical location of brain metastasis, and requiring patients with new asymptomatic metastasis to receive radiotherapy/surgery before enrolling in this study, will be determined per investigator's medical judgement and consultation.
4. Active autoimmune diseases or history of autoimmune diseases that may relapse.

   Note: Patients with the following diseases are not excluded and may proceed to further screening:
   1. Controlled Type I diabetes
   2. Hypothyroidism (provided it is managed with hormone replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors
5. Any active malignancy ≤2 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
6. Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before first dose of study drug.

   Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:
   1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
   3. Short course (≤7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
7. With uncontrolled diabetes or >Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥Grade 3 hypoalbuminemia ≤14 days before first dose of study drug.
8. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.; an assessment of pulmonary function will be conducted at screening (see Section 7.1.4)
9. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.

   * Severe infections within 4 weeks before or first dose of study drug, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
   * Received therapeutic oral or intravenous antibiotics within 2 weeks before first cycle of study drug
10. A known history of HIV infection.
11. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is >500 IU/mL or patients with active hepatitis C virus (HCV) should be excluded.

    Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA <500 IU/mL), and cured hepatitis C patients can be enrolled.
12. Any major surgical procedure requiring general anesthesia ≤28 days before first dose of study drug.
13. Prior allogeneic stem cell transplantation or organ transplantation.
14. Any of the following cardiovascular risk factors:

    1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤28 days before first dose of study drug
    2. Pulmonary embolism ≤28 days before first dose of study drug
    3. Any history of acute myocardial infarction ≤6 months before first dose of study drug
    4. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV ≤6 months before first dose of study drug (Appendix 6)
    5. Any event of ventricular arrhythmia ≥Grade 2 in severity ≤6 months before first dose of study drug
    6. Any history of cerebrovascular accident ≤6 months before first dose of study drug
    7. Uncontrolled hypertension: systolic pressure ≥160 mmHg or diastolic pressure ≥100 mmHg despite anti-hypertension medications ≤28 days before first dose of drug
    8. Any episode of syncope or seizure ≤28 days before first dose of study drug
15. A history of severe hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
16. Has received any chemotherapy, immunotherapy (e.g., interleukin, interferon, thymosin) or any investigational therapies within 28 days or 5 half-lives (whichever is shorter) of the first study drug administration.
17. Has received any herbal medicine used to control cancer within 14 days of the first study drug administration.
18. Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy and specific laboratory abnormalities).
19. Was administered a live vaccine ≤4 weeks before first dose of study drug. Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. COVID-19 vaccines are allowed if not live vaccines. Intranasal vaccines are live vaccines, and are not allowed.
20. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct.
21. Concurrent participation in another therapeutic clinical study.
22. Has QT corrected (QTc) interval (corrected by Fridericia's method) >470 msec (if applicable).

    Note: If any patient has QTc interval >450 msec on initial ECG, follow up ECG will be performed [in triplicate] to exclude result
23. Received radiation therapy within 14 days prior to randomization.
24. Total lifetime anthracycline load exceeding 360 mg/m2 doxorubicin or equivalent.
25. Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease (with exception of subjects with Gilbert's Syndrome, asymptomatic gall stones, liver metastases, or stable chronic liver disease per investigator assessment).
26. Females who are breastfeeding or pregnant, and females and males planning a pregnancy.
27. With the following disease-related risk factors:

    1. Clinically significant bleeding (≥Grade 3) from the gastrointestinal (GI) tract within 4 weeks prior to randomization
    2. Clinically significant bowel obstruction (≥Grade 3)
28. Accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to randomization. Receipt of diuretic drugs for other reasons is acceptable

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG RHA, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea